CLINICAL TRIAL: NCT00693719
Title: A Phase II Study: Irinotecan and Etoposide as Treatment for Refractory, Metastatic Breast Cancer
Brief Title: Irinotecan and Etoposide in Treating Patients With Recurrent, Locally Advanced, or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0327-04; P30CA016672 (NIH); UARIZ-BIO07046 (Other: University of Arizona); UARIZ-143 (Other: University of Arizona); PFIZER-GA59608L (Other Grant/Funding Number: Pfizer); UARIZ-P18089 (Other: University of Arizona)
Record Dates: First submitted 2008-06-06; First posted 2008-06-09 (Estimated); Results first posted 2013-08-21 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Etoposide; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etoposide and Irinotecan hydrochloride (Experimental): Irinotecan 100 mg/m2 IV days 1 and 15. Etoposide 50 mg PO x14 days followed by 2 weeks off.
  Interventions: Drug: Etoposide; Drug: Irinotecan hydrochloride

INTERVENTIONS:
Drug: Etoposide — 50 mg PO x14 days followed by 2 weeks off, 28 day/Cycle
  Other Names: Vepesid
Drug: Irinotecan hydrochloride — Irinotecan 100 mg/m2 IV days 1 and 15, 28 day/Cycle
  Other Names: Irinotecan hydrochloride trihydrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving irinotecan together with etoposide works in treating patients with recurrent, locally advanced, or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the response rate, as assessed by RECIST criteria, in patients with recurrent locally advanced or metastatic breast cancer treated with irinotecan hydrochloride and etoposide after prior exposure to anthracycline, taxane, and capecitabine therapy.

Secondary

* To determine the median time to progression in these patients.
* To determine the response duration and survival in these patients.
* To measure the type and rate of grade 3 or greater toxicity of this treatment regimen in these patients.

OUTLINE: Patients receive irinotecan hydrochloride IV on days 1 and 15 and oral etoposide on days 1-14. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.

After completion of study therapy, patients are followed every 3 months for 3 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of locally advanced or metastatic breast cancer

  * Recurrent, refractory or progressive disease after receiving prior anthracycline, taxane, and capecitabine therapy

    * Prior anthracycline and taxane therapy may have been as neoadjuvant, or adjuvant therapy if disease progression is documented within a year of completing that agent
    * Received prior capecitabine therapy for metastatic or recurrent disease
* Measurable disease

  * Bone metastases requires other disease present that can be measured
* No brain metastases, unless documented to be controlled post-completion of local therapy (surgery and/or radiation therapy) for at least 4 weeks
* No meningeal carcinomatosis
* No malignant effusion as the only site of disease recurrence
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Performance status of 0-2
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 40 mL/min
* Hemoglobin ≥ 10 g/dL
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal or hyperbilirubinemia < grade 1 (unless due to Gilbert syndrome with elevated total but normal levels of conjugated bilirubin)
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other non-breast malignancy, except nonmelanoma skin cancer
* No other serious underlying medical condition, that in the opinion of the treating physician, would make study protocol unreasonably hazardous for the patient or would preclude the patient's ability to comply with the study protocol

PRIOR CONCURRENT THERAPY:

* See Disease Characteristic
* Recovered from all prior chemotherapy or radiotherapy to NCI CTC grade ≤ 1
* Unlimited documented prior chemotherapy regimens allowed
* No prior irinotecan hydrochloride or etoposide
* No Hypericum perforatum (St. John's wort) 14 days prior to, during, or 7 days after completion of study therapy
* At least 7 days since prior and no concurrent phenytoin, carbamazepine, phenobarbital, or any other enzyme-inducing anticonvulsant drug (EIACD)
* No concurrent aprepitant

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-08; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B. Livingston, MD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona, United States

REFERENCES:
- [Derived] Segar JM, Reed D, Stopeck A, Livingston RB, Chalasani P. A Phase II Study of Irinotecan and Etoposide as Treatment for Refractory Metastatic Breast Cancer. Oncologist. 2019 Dec;24(12):1512-e1267. doi: 10.1634/theoncologist.2019-0516. Epub 2019 Aug 5. PMID 31383812

RESULTS

PARTICIPANT FLOW:
Groups:
- Etoposide/Irinotecan: Irinotecan hydrochloride : Irinotecan 100 mg/m2 IV days 1 and 15, 28 day/Cycle
  Etoposide : 50 mg PO x14 days followed by 2 weeks off, 28 day/Cycle
Period: Overall Study
Arm/Group | Etoposide/Irinotecan
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Etoposide/Irinotecan
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.68 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Measured time from the start of treatment to the time the patient is first recorded as having disease progression or dies. If no progression or death while being followed via tumor assessment, censored at last date known alive, assesed up to 13 months
Measure: Median (Standard Error); unit: Days
Arm/Group | Etoposide/Irinotecan
Number analyzed (Participants) | 31
Days | 149 (33.83)

2. Secondary Outcome: Overall Survival
Description: Still alive for a certain period of time after they were diagnosed with or started treatment
Time Frame: Measured from the start of protocol therapy until the date of death from any cause or will be censored at the date the patient was last known to be alive, assesed up to 13 months
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Etoposide/Irinotecan
Number analyzed (Participants) | 31
Days | 149 [82.703 to 215.297]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at the end of each 28-day cycle of treatment
Arm/Group | Etoposide/Irinotecan
Serious Adverse Events (participants affected / at risk) | 4/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoposide/Irinotecan (N=31)
Pain (Gastrointestinal disorders) | 2 (3)
Dehydration (Gastrointestinal disorders) | 1 (1)
Dyspnea (General disorders) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etoposide/Irinotecan (N=31)
Nausea (Gastrointestinal disorders) | 22 (36)
Diarrhea (Gastrointestinal disorders) | 13 (33)
Vomiting (Gastrointestinal disorders) | 10 (18)
Anorexia (Gastrointestinal disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 6 (7)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 6 (6)
Ascites (non-malignant) (Gastrointestinal disorders) | 4 (4)
Dehydration (Gastrointestinal disorders) | 4 (5)
Distension/bloating, abdominal (Gastrointestinal disorders) | 4 (7)
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 4 (11)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3 (3)
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 3 (4)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 25 (78)
Hemoglobin (Blood and lymphatic system disorders) | 21 (74)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 19 (77)
Platelets (Blood and lymphatic system disorders) | 11 (34)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 15 (40)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 13 (34)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 12 (19)
Alkaline phosphatase (Metabolism and nutrition disorders) | 11 (18)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 11 (23)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 9 (17)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 6 (7)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5 (11)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (13)
Pain - Other (Specify, __) (General disorders) | 10 (15)
Pain - Abdomen NOS (General disorders) | 8 (17)
Pain - Bone (General disorders) | 7 (9)
Pain - Throat/pharynx/larynx (General disorders) | 5 (7)
Pain - Back (General disorders) | 4 (5)
Pain - Pelvis (General disorders) | 4 (6)
Pain - Chest/thorax NOS (General disorders) | 2 (2)
Pain - Extremity-limb (General disorders) | 2 (4)
Pain - Head/headache (General disorders) | 2 (2)
Pain - Joint (General disorders) | 2 (2)
Pain- Rectum (General disorders) | 2 (2)
Pain - Stomach (General disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 14 (21)
Weight loss (General disorders) | 4 (4)
Insomnia (General disorders) | 3 (3)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (3)
Sweating (diaphoresis) (General disorders) | 2 (2)
Dizziness (General disorders) | 6 (6)
Confusion (General disorders) | 3 (4)
Neuropathy: sensory (General disorders) | 3 (3)
Mood alteration - Anxiety (Psychiatric disorders) | 2 (5)
Neurology - Other (Specify, __) (General disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 10 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 2 (2)
Infection - Other (Specify, __) (Infections and infestations) | 2 (2)
Infection with unknown ANC - Upper airway NOS (Infections and infestations) | 2 (2)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 4 (5)
Flushing (Skin and subcutaneous tissue disorders) | 3 (5)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (5)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 (2)
Edema: limb (Blood and lymphatic system disorders) | 5 (6)
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 2 (3)
Hot flashes/flushes (Endocrine disorders) | 3 (3)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (2)
Cardiopulmonary arrest, cause unknown (non-fatal) (Cardiac disorders) | 2 (3)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes